CLINICAL TRIAL: NCT05811481
Title: Clinical Research and Laboratory Animal Ethics Committee of the First Affiliated Hospital of Sun Yat-sen University
Brief Title: Regorafenib Alone or in Combined With Transcatheter Arterial ChEmoembolization in Treatment of Advanced Hepatocellular Carcinoma After First Line Targeted Therapy
Acronym: ROSE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: WenBo Guo (Other)
Responsible Party: Sponsor-Investigator, WenBo Guo, professor, First Affiliated Hospital, Sun Yat-Sen University
Organization: First Affiliated Hospital, Sun Yat-Sen University (Other)
Other Study IDs: [2022]662
Record Dates: First submitted 2023-03-26; First posted 2023-04-13 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Hepatocellular Carcinoma; Transcatheter Arterial ChEmoembolization; Regorafenib
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — regorafenib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Two treatment groups: Regorafenib + TACE
  Interventions: Procedure: TACE; Drug: Regorafenib
- Treatment ate group: Regorafinib
  Interventions: Drug: Regorafenib

INTERVENTIONS:
Procedure: TACE — Transcatheter Arterial Chemoembolization
  Groups: Two treatment groups
Drug: Regorafenib — Regorafenib alone

SUMMARY:
. 1 Clarify the difference in efficacy of regofinib combined with TACE compared with second-line treatment of advanced liver cancer; 2. To evaluate the safety and prognostic imaging factors of regorofenib in advanced second-line therapy; 3, to explore whether it is necessary to increase the treatment of TACE in the second-line treatment of advanced HCC.

ELIGIBILITY:
Inclusion Criteria:

( - ) After pathological / clinical diagnosis of hepatocellular carcinoma or radical resection of hepatocellular carcinoma; ( - ) CNLC Ⅲa Patients with intrahepatic recurrence before (including a); ( - ) Previous failure of first-line systemic treatment; ( - ) Age: 18-75 years old; ( - ) Child-Pugh 7 points; ( - ) ECOG PS Grade 0-2; ( - ) At least one measurable lesion in the liver.

Exclusion Criteria:

( - ) Known hepatobiliary tubular cell carcinoma and mixed cell carcinoma and fibrolamellar cell carcinoma; ( - ) Previous (within 5 years) or concurrent other incurable malignant tumors; ( - ) Having received local treatment, systemic chemotherapy, radiotherapy other than TACE during the first-line systemic treatment; ( - ) During the second-line systemic treatment, I also received local treatment, systemic chemotherapy, radiotherapy other than TACE; ( - ) Serious uncontrollable systemic and other systemic diseases, such as uremia, cardiovascular and cerebrovascular accidents; ( - ) Allergy to any drug included in the study; ( - ) Pregnant or lactating women;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hepatocellular carcinoma
Sampling Method: Probability Sample
Enrollment: 192 (Estimated)
Dates: Start 2022-12-27 (Actual); Primary Completion 2024-12-27 (Estimated); Study Completion 2025-12-27 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 2022.12.27-2025.09.30
  defined as the time between the start of second-line treatment and the end of follow-up / death.

SECONDARY OUTCOMES:
Progression-free survival for the first subsequent treatment PFS 2 | 2022.12.27-2025.09.30
  defined as the time of second-line treatment initiation to the date of radiological progression or death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- FirstSunYetSen, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
Regorafenib Alone or in Combined with Transcatheter Arterial ChEmoembolization in Treatment of Advanced Hepatocellular Carcinoma after First Line Targeted Therapy